CLINICAL TRIAL: NCT02494609
Title: A Two-way Study to Evaluate the Potential Pharmacokinetic Interactions Between Sotagliflozin (LX4211) and Ortho-Cyclen®, an Oral Contraceptive Containing Norgestimate and Ethinyl Estradiol, in Healthy Premenopausal Women
Brief Title: Oral Contraceptive DDI Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LX4211.1-120-NRM; LX4211.120 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): once daily dosing for 7 days, followed by 7-day washout
  Interventions: Drug: sotagliflozin
- Treatment B (Experimental): once daily dosing for 28 days
  Interventions: Drug: oral contraceptive
- Treatment C (Experimental): once daily dosing for 14 days of oral contraceptive, followed by coadministration with sotagliflozin once daily for 7 days
  Interventions: Drug: oral contraceptive + sotagliflozin

INTERVENTIONS:
Drug: sotagliflozin — 400 mg sotagliflozin
  Arms: Treatment A
Drug: oral contraceptive — 0.25 mg norgestimate/0.035 mg ethinyl estradiol
  Arms: Treatment B
Drug: oral contraceptive + sotagliflozin — 0.25 mg norgestimate/0.035 mg ethinyl estradiol + 400 mg sotagliflozin
  Arms: Treatment C

SUMMARY:
A Two-way Study to Evaluate the Potential Pharmacokinetic Interactions Between Sotagliflozin (LX4211) and an Oral Contraceptive Containing Norgestimate and Ethinyl Estradiol, in Healthy Premenopausal Women.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females with a body mass index (BMI) between 18 and 32 kg/m2 (inclusive)
* Have not received any oral contraceptives during the Screening period or for at least 15 days prior to the first dose of Period 1

Exclusion Criteria:

* History of any contraindications to the combined oral contraceptive tablet including thrombosis and the history of any thromboembolic disease, recurrent jaundice, acute or chronic liver disease, hormonally-induced migraines, undiagnosed vaginal bleeding, significant hyperlipidemia, and mammary, endometrial, or hepatic carcinoma (known or suspected)
* Prior exposure to sotagliflozin (LX4211)
* History of any clinically relevant psychiatric, renal, hepatic, pancreatic, endocrine, cardiovascular, neurological, hematological, or GI abnormality
* Concurrent conditions that could interfere with safety and/or tolerability measurements
* Women who are breastfeeding or are planning to become pregnant during the study
* Positive serum pregnancy test
* Have taken injectable contraceptives or hormonal intrauterine devices within 12 months prior to the first dose of Period 1 or topical controlled delivery contraceptives (patch) for 3 months prior to the first dose of Period 1

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of sotaglifozin to evaluate protocol specified PK parameters | Day 6 to Day 8, Day 55 to Day 57, Day 62 to Day 64
Plasma concentration of norgestimate/ethinyl estradiol to evaluate protocol specified PK parameters | Day 55 to Day 57, Day 62 to Day 64

SECONDARY OUTCOMES:
Number of treatment emergent adverse events | Day 1 to Day 70

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Lexicon Investigational Site, Evansville, Indiana
  - Lexicon Investigational Site, Dallas, Texas